CLINICAL TRIAL: NCT06150924
Title: A Randomized, Crossover, Double Blind, Placebo Controlled, Phase 2 Study to Evaluate the Efficacy and Safety of Lorundrostat in Addition to Sodium-Glucose Cotransporter-2 Inhibitors, in Adults With Hypertension and Chronic Kidney Disease With Albuminuria
Brief Title: Efficacy and Safety of Lorundrostat in Addition to Sodium-Glucose Cotransporter-2 Inhibitors (SGLT2i) in Subjects With Hypertension and Chronic Kidney Disease (CKD) With Albuminuria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mineralys Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MLS-101-206
Record Dates: First submitted 2023-11-17; First posted 2023-11-29 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Chronic Kidney Disease
Keywords: Albuminuria; Arterial hypertension; Hypertension; Proteinuria; Diabetic nephropathy; Chronic Kidney Disease; Aldosterone Synthase Inhibitor
MeSH Terms: conditions — Renal Insufficiency, Chronic; Albuminuria; Hypertension; Proteinuria; Diabetic Nephropathies

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Experimental)
  Interventions: Drug: Lorundrostat 25mg+SGLT2i QD, Washout, Placebo+SGLT2i QD
- Cohort 2 (Experimental)
  Interventions: Drug: Placebo QD + SGLT2i QD, Washout, Lorundrostat 25mg+SGLT2i QD

INTERVENTIONS:
Drug: Lorundrostat 25mg+SGLT2i QD, Washout, Placebo+SGLT2i QD — Period 1 - Lorundrostat 25mg QD + SGLT2i QD 4 weeks; Washout - Placebo QD + SGLT2i QD 4 weeks; Period 2 - Placebo QD + SGLT2i QD 4 weeks
  Arms: Cohort 1
Drug: Placebo QD + SGLT2i QD, Washout, Lorundrostat 25mg+SGLT2i QD — Period 1 - Placebo QD + SGLT2i QD 4 weeks; Washout - Placebo QD + SGLT2i QD 4 weeks; Period 2 - Lorundrostat 25mg + SGLT2i QD 4 weeks
  Arms: Cohort 2

SUMMARY:
This is a randomized, double-blind (DB), placebo controlled, crossover study with a two-period, two-sequence (2x2) design evaluating the efficacy and safety of 25 mg QD lorundrostat (an aldosterone synthase inhibitor [ASI]) in addition to a SGLT2i for the treatment of hypertension in subjects with CKD and albuminuria while receiving stable treatment with an Angiotensin-converting enzyme inhibitor (ACEi) or an Angiotensin receptor blocker (ARB). Subjects will be at least 18 years old with hypertension, and mild to severe CKD with albuminuria at the Screening Visit.

DETAILED DESCRIPTION:
The study consists of up to a 2-week Screening period, a 2-week run-in period where subjects will either begin study provided dapagliflozin 10 mg or continue on their regularly prescribed SGLT2i, and two DB 4-week treatment periods separated by a 4-week washout period. Subjects will be randomized (1:1) to two treatment sequences: lorundrostat-placebo (LP) and placebo-lorundrostat (PL).

ELIGIBILITY:
Major Inclusion Criteria:

1. At Screening, UACR of 200-5000 mg/g, inclusive, in first morning urine void
2. At Screening, eGFRs of ≥30 mL/min/1.73 m2
3. At Screening, AOBP SBP of 135-180 mmHg, inclusive
4. On a stable treatment with an ACEi or ARB for at least 2 months prior to Screening
5. At Screening, body mass index (BMI) of >18 kg/m2

Major Exclusion Criteria:

1. Subjects with known hypersensitivity to lorundrostat or any of its respective excipients
2. Subjects with known hypersensitivity to dapagliflozin or any of its respective excipients (subjects beginning dapagliflozin only)
3. At Screening, serum potassium >5.0 mmol/L
4. History of clinically significant hyponatremia within 1 year prior to Screening
5. Use of epithelial sodium channel (ENaC) inhibitors or Mineralocorticoid receptor antagonist (MRAs), including, but not limited to amiloride, triamterene, spironolactone, eplerenone, finerenone, from 4 weeks prior to the Screening Visit and during study participation. With the exception of MRAs in primary aldosteronism
6. Medical history of kidney disease related to autoimmune diseases (lupus, anti-neutrophil cytoplasmic antibody [ANCA] vasculitis), multiple myeloma or other known paraproteins, infiltrative diseases of the kidney, obstructive nephropathy, cystic kidney diseases, and renal transplantation
7. Medical history of advanced liver disease, including cirrhosis
8. Medical history of active autoimmune disease or recent (within 30 days) or anticipated need for immunosuppressive therapy
9. Diabetes mellitus with a glycosylated hemoglobin (HbA1c) >10% (>86 mmol/mol) at Screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-12-14 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-04-23 (Actual)

PRIMARY OUTCOMES:
Placebo-adjusted change from baseline in automated office blood pressure (AOBP) systolic blood pressure (SBP) at Week 4 | baseline to Week 4
Incidence and severity of adverse events (AEs) | baseline to Week 14

OTHER OUTCOMES:
Placebo-adjusted percent change from baseline in 24-hour urine albumin at Study Week 4 | baseline to Study Week 4
Placebo-adjusted change from baseline in AOBP diastolic blood pressure (DBP) at Study Week 4 | Study Week 4
Change from baseline in AOBP SBP at Study Week 4 lorundrostat treatment periods | Study Week 4
Percent change from baseline in 24-hour urine albumin at Study Week 4 in lorundrostat treatment periods | baseline to Study Week 4
Placebo-adjusted percent change from baseline in 24-hour urine protein Study Week 4 | baseline to Study Week 4
Placebo-adjusted percent change from baseline in urine albumin to creatinine ratio (UACR) at Study Week 4 | baseline to Study Week 4
Change in biomarkers from baseline to Study Week 4 in lorundrostat treatment periods | baseline to Study Week 4
Placebo-adjusted percent change in estimated glomerular filtration rate (eGFR) from baseline to Study Week 4 | baseline to Study Week 4
Percent change in eGFR from Study Week 4 to Study Week 8 | Study Week 4 to Study Week 8

CONTACTS AND LOCATIONS:
Locations (44):
- United States (44):
  - Arizona Kidney Disease & Hypertension Centers (AKDHC) - Thunderbird Office, Glendale, Arizona
  - Arizona Kidney Disease & Hypertension Centers (AKDHC) - Thomas Office, Phoenix, Arizona
  - Balboa Nephrology Medical Group, Inc. (BNMG) - California Institute of Renal Research (CIRR) - Chula Vista, Chula Vista, California
  - Balboa Nephrology Medical Group, Inc. (BNMG) - El Centro, El Centro, California
  - Amicis Research Center - Granada Hills, Granada Hills, California
  - Balboa Nephrology Medical Group, Inc. (Bnmg) - La Mesa, La Mesa, California
  - Academic Medical Research Institute (AMRI) - Los Angeles, Los Angeles, California
  - Amicis Research Center, Northridge, California
  - Amicis Research Center - Vacaville, Vacaville, California
  - Colorado Kidney Care (Denver Nephrology) - Denver Office, Denver, Colorado
  - Qway Research, Coconut Grove, Florida
  - Indago Research and Health Center, Hialeah, Florida
  - Elixia Pines, LLC, Hollywood, Florida
  - Elixia Central Florida, LLC, Orlando, Florida
  - Infigo Clinical Research, Llc, Sanford, Florida
  - Genesis Clinical Research - Tampa, Tampa, Florida
  - Palm Beach Diabetes and Endocrine Specialists, PA (PBDES) - West Palm Beach Office, West Palm Beach, Florida
  - American Clinical Trials Llc, Acworth, Georgia
  - Nephrology of the Golden Isles - Brunswick, Brunswick, Georgia
  - ClinCept, LLC, Columbus, Georgia
  - Georgia Nephrology, Llc, Lawrenceville, Georgia
  - Nephrology Associates of Kentuckiana, PSC (NAK), Louisville, Kentucky
  - Lcms Health University Medical Center New Orleans, New Orleans, Louisiana
  - Northwest Louisiana Nephrology, Llc - Shreveport, Shreveport, Louisiana
  - Tufts University School of Medicine (Tusm) - Tufts Medical Center (Tmc) (Tufts-New England Medical Center), Boston, Massachusetts
  - Elixia MKC, LLC, Pontiac, Michigan
  - Kansas City Kidney Consultants (Arms, Dodge, Robinson, Wilber & Crouch, Inc.) - Kansas City, Kansas City, Missouri
  - Seacoast Kidney & Hypertension Specialists - Portsmouth Office, Portsmouth, New Hampshire
  - Suny Downstate Medical Center - Parkside Dialysis Center, Brooklyn, New York
  - Nephrology Associates, PC, Fresh Meadows, New York
  - Nephrology Associates, Fresh Meadows, New York
  - Triad Internal Medicine, Asheboro, North Carolina
  - Nephrology Associates, Pllc - Winston-Salem, Winston-Salem, North Carolina
  - Nephrology Consultants - Oklahoma City, Oklahoma City, Oklahoma
  - Columbia Nephrology, Columbia, South Carolina
  - Southeast Renal Research Institute, Chattanooga, Tennessee
  - Dallas Nephrology Associates (Dna) - Renal Disease Research Institute (Rdri), Dallas, Texas
  - Liberty Research Center, Dallas, Texas
  - R&H Clinical Research, Katy, Texas
  - E T Nephrology Associates - Lufkin, Lufkin, Texas
  - Prx Research, Mesquite, Texas
  - Gamma Medical Research, Inc, Mission, Texas
  - Chrysalis Clinical Research (CCR), St. George, Utah
  - Mendez Center for Clinical Research, LLC, Woodbridge, Virginia

IPD SHARING:
Plan to Share IPD: No